CLINICAL TRIAL: NCT02440269
Title: The Effect of Circadian Rhythms on Norctrend Index in Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lu KZ (Other)
Responsible Party: Sponsor-Investigator, Lu KZ, Director, Head of anesthesiology, Southwest Hospital, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Other Study IDs: narcotrend
Record Dates: First submitted 2015-05-03; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Patients Needed Surgery and Anesthesia; Except on the Head or Facial Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A：day: the patients who receive surgery and anesthesia during 8:00 am to 6:00 pm
- B：night: the patients who receive surgery and anesthesia during 10:00 pm to 5:00 am next day

SUMMARY:
The purpose of this study is to determine whether the Circadian Rhythms effects on the Norctrend Index in Anesthesia.

DETAILED DESCRIPTION:
It has been reported that circadian rhythm has many aspects of influence on human body. But little is knew about the circadian rhythm affect on Narcotrend index (made in Germany) in total intravenous anesthesia .The investigators' study is to find the relationship between them.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists（ASA） Ⅰ - Ⅱ;
* ability to compliance the research plan;
* volunteered and signed for the study ;
* receive surgery and general anesthesia

Exclusion Criteria:

* ASA>Ⅱ;
* Head or facial surgery
* can't collaborate;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who receive surgery and general anesthesia
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
narcotrend index | during operation time
  the narcotrend index we recorded during the surgery and anesthesia in appropriate depth of anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Southwest Hospital Third Military Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Shen JH, Ye M, Chen Q, Chen Y, Zhao HL, Khan A, Yi B, Ning JL, Lu KZ, Gu JT. Effects of circadian rhythm on Narcotrend index and target-controlled infusion concentration of propofol anesthesia. BMC Anesthesiol. 2021 Sep 6;21(1):215. doi: 10.1186/s12871-021-01445-z. PMID 34488646